CLINICAL TRIAL: NCT01739933
Title: Altering Sedation Paradigms to Improve Brain Injury and Survival in Severe Sepsis
Brief Title: The MENDS2 Study, Maximizing the Efficacy of Sedation and Reducing Neurological Dysfunction and Mortality in Septic Patients With Acute Respiratory Failure
Acronym: MENDS2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Pratik Pandharipande, Professor of Anesthesiology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R01HL111111 (NIH); 121380 (Other: Vanderbilt University Institutional Review Board)
Record Dates: First submitted 2012-11-28; First posted 2012-12-04 (Estimated); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Sepsis; Delirium; Impaired Cognition
Keywords: Delirium; Delirium/coma-free days; Long term cognitive impairment; Sedation; Intensive care; Mechanical Ventilation; Dexmedetomidine; Propofol; Coma-free days; Sepsis; Organ dysfunction; Acute Respiratory Distress; Markers of inflammation
MeSH Terms: conditions — Sepsis; Delirium; Cognition Disorders; Acute Lung Injury | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Active Comparator): Route and Concentration. The study drug will be administered intravenously (IV) by continuous infusion at concentrations of 5 mcg/mL dexmedetomidine. Patients will only receive study drug while in the ICU and on mechanical ventilation, and thus will be monitored with continuous telemetry as per usual ICU practice.
  Dosing Range. Study drug dose will be titrated in a double-blind manner according to clinical effect to achieve a "goal" or "target" Richmond Agitation Sedation Score set by the managing clinical team. For patients in the dexmedetomidine group, dose will range from 0.15-1.5 mcg/kg/hr.
  Interventions: Drug: Dexmedetomidine
- Propofol (Active Comparator): Route and Concentration. The study drug will be administered intravenously (IV) by continuous infusion at concentrations of 10 mg/mL propofol. Patients will only receive study drug while in the ICU and on mechanical ventilation, and thus will be monitored with continuous telemetry as per usual ICU practice.
  Dosing Range. Study drug dose will be titrated in a double-blind manner according to clinical effect to achieve a "goal" or "target" Richmond Agitation Sedation Score set by the managing clinical team. For patients in the propofol group, dose will range from 5-50 mcg/kg/min.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — For patients in the dexmedetomidine group, dose will range from 0.15-1.5 mcg/kg/hr. For example, a 70 kg patient would receive 10.5 mL of study drug per hour, which would provide 0.75 mcg/kg/hr of dexmedetomidine. This dose range have been selected after literature review and discussions with critical care practitioners, investigational pharmacists, and the MENDS2 study steering committee.
  Other Names: Precedex; Dexdor
  Arms: Dexmedetomidine
Drug: Propofol — For patients in the propofol group, dose will range from 5-50 mcg/kg/min. For example, a 70 kg patient would receive 10.5 mL of study drug per hour, which would provide 25 mcg/kg/min of propofol. This dose range has been selected after literature review and discussions with critical care practitioners, investigational pharmacists, and the MENDS2 study steering committee.
  Other Names: Diprivan
  Arms: Propofol

SUMMARY:
Ventilated ICU patients frequently have sepsis and the majority have delirium, a form of brain dysfunction that is an independent predictor of increased risk of dying, length of stay, costs, and prolonged cognitive impairment in survivors. Universally prescribed sedative medications-the GABA-ergic benzodiazepines-worsen this brain organ dysfunction. The available alternative sedation regimens, the shorter acting GABA-ergic propofol, and the alpha2 agonist, dexmedetomidine, have both been shown to be superior to benzodiazepines, and yet are different with regard to their effects on innate immunity, bacterial clearance, apoptosis, cognition and delirium. The MENDS2 study will compare propofol and dexmedetomidine, and determine the best sedative medication to reduce delirium and improve survival and long-term brain function in our most vulnerable patients- the ventilated septic patient.

DETAILED DESCRIPTION:
The need for mechanical ventilation (MV) secondary to sepsis is the leading cause of admission to the intensive care unit, often necessitating sedation for patient safety and comfort. Recently, we have learned that these sedative medications contribute to iatrogenic injury, such as prolonging ventilator time and ICU length of stay and exacerbating acute brain dysfunction. This acute brain dysfunction, manifested as delirium and coma, occurs in 50%-70% of MV septic patients and is a significant contributor not only to death but also to functional and cognitive decline, which can persist for years after recovery of lung and other organ function, levying significant costs to patients and society. Despite advances in the management of acute respiratory failure and sepsis, few clinical trials have examined the effects that supportive therapies, like sedation, may have on both short- and long-term outcomes in this vulnerable population. The gamma-aminobutyric acid (GABA)-ergic benzodiazepines, in particular, have been shown to increase brain dysfunction, promote infection, and prolong MV. Therefore, the short-acting GABA-ergic sedative propofol and the alpha2 agonist dexmedetomidine are becoming widely used to sedate septic MV patients. There are only a few randomized trials, however, to guide clinicians when selecting between these and other sedatives, and none have explored the mechanisms underlying the differences in outcomes, though some data indicate that GABA-ergic and alpha2 agonist agents have very different effects on innate immunity, apoptosis, arousability, and respiratory drive. In early animal and human studies, dexmedetomidine had more anti-inflammatory effects than the GABA-ergic agents; dexmedetomidine improved bacterial clearance, whereas propofol impaired it. In addition, sedation with dexmedetomidine instead of benzodiazepines reduces delirium by 20%-30% and improves arousability, cognition, and attentiveness in ventilated patients. Alpha2 agonists induce unconsciousness at the brainstem-more akin to natural sleep-which may improve autonomic function and immunity. All these factors converge to suggest that sedation with an alpha2 agonist rather than a GABAergic agent may improve outcomes, including brain function, MV, and survival, for septic MV patients. We therefore propose the MENDS2 (Maximizing the Efficacy of Sedation and Reducing Neurological Dysfunction and Mortality in Septic Patients with Acute Respiratory Failure) study, in which we will test the hypotheses that sedation of MV severely septic patients with an alpha2 agonist (dexmedetomidine) rather than a GABAergic agent (propofol) will (Aim 1A) increase days alive without delirium or coma, (Aim 1B) increase ventilator-free days, (Aim 2A) improve 90-day survival, (Aim 2B) decrease long-term cognitive impairment, and (Aim 3) reduce the pro-inflammatory cytokine cascade following sepsis. We will randomize 420 ventilated, severely septic patients requiring goal-directed sedation with dexmedetomidine or propofol, giving the study 85% power to detect a difference of 1.5 delirium/coma-free days and an absolute difference in mortality of 12% between the two groups.

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients will be eligible for inclusion in the MENDS2 study if they are: [1] adult patients (≥18 years old) [2] in a medical and/or surgical ICU and [3] on MV and requiring sedation and [4] have suspected or known infection

Exclusion Criteria:

Patients will be excluded (i.e., not consented) for any of the following reasons:

1. Rapidly resolving organ failure, indicated by planned immediate discontinuation of MV, at time of screening for study enrollment
2. Pregnant or breastfeeding
3. Severe dementia or neurodegenerative disease, defined as either impairment that prevents the patient from living independently at baseline or IQCODE >4.5, measured using a patient's qualified surrogate. This exclusion also pertains to mental illnesses requiring long-term institutionalization, acquired or congenital mental retardation, severe neuromuscular disorders, Parkinson's disease, and Huntington's disease. It also excludes patients in coma or with severe deficits due to structural brain diseases such as stroke, intracranial hemorrhage, cranial trauma, malignancy, anoxic brain injury, or cerebral edema.
4. History of 2nd or 3rd degree heart block, bradycardia < 50 beats/minute, pacemaker for bradyarrythmias or uncompensated shock.If patient has a pacemaker for bradyarrythmias, then patient does not meet this exclusion criterion and may be enrolled.
5. Benzodiazepine dependency or history of alcohol dependency based on the medical team's decision to institute a specific treatment plan involving benzodiazepines (either as continuous infusions or intermittent intravenous boluses) for this dependency.
6. Active seizures during this ICU admission being treated with intravenous benzodiazepines.
7. Expected death within 24 hours of enrollment or lack of commitment to aggressive treatment by family/medical team (e.g., likely to withdraw life support measures within 24 hrs of screening)
8. Inability to understand English or deafness or vision loss that will preclude delirium evaluation. The inability to understand English (for example in Spanish-only or Mandarin-only speaking patients) will not result in exclusion at centers where the research staff is proficient and/or translation services are actively available in that particular language; these patients will not be followed in the long-term follow-up phase of the trial since the testing materials are primarily available only in English. Patients with laryngectomies and those with hearing deficits are eligible for enrollment if their medical condition permits them to communicate with research staff.
9. Inability to obtain informed consent from an authorized representative within 48 hours of meeting all inclusion criteria, i.e., developing sepsis and qualifying organ dysfunction criteria for the following reasons:

   1. Attending physician refusal.
   2. Patient and/or surrogate refusal.
   3. Patient unable to consent and no surrogate available.
   4. 48-hour period of eligibility was exceeded before the patient was screened.
10. Prisoners.
11. Medical team following patient unwilling to use the sedation regimens.
12. Documented allergy to propofol or dexmedetomidine.
13. Current enrollment in a study that does not allow co-enrollment or that uses delirium as a primary outcome.
14. Patients who are on muscle relaxant infusions at time of screening with plans to maintain paralysis >48 hours.
15. Greater than 96 hours on mechanical ventilation prior to meeting all inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2013-05-15 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pratik P. Pandharipande, MD, MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (11):
- United States (11):
  - University of California, San Francisco, San Francisco, California
  - Baton Rouge General Medical Center and Our Lady of The Lakes Regional Medical Center, Baton Rouge, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Mission Hospital, Asheville, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Health Harris Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Hughes CG, Mailloux PT, Devlin JW, Swan JT, Sanders RD, Anzueto A, Jackson JC, Hoskins AS, Pun BT, Orun OM, Raman R, Stollings JL, Kiehl AL, Duprey MS, Bui LN, O'Neal HR Jr, Snyder A, Gropper MA, Guntupalli KK, Stashenko GJ, Patel MB, Brummel NE, Girard TD, Dittus RS, Bernard GR, Ely EW, Pandharipande PP; MENDS2 Study Investigators. Dexmedetomidine or Propofol for Sedation in Mechanically Ventilated Adults with Sepsis. N Engl J Med. 2021 Apr 15;384(15):1424-1436. doi: 10.1056/NEJMoa2024922. Epub 2021 Feb 2. PMID 33528922
- [Derived] Chandrasekhar R, Hughes CG, Pun BT, Orun OM, Ely EW, Pandharipande PP. Statistical analysis plan for the Maximizing the Efficacy of Sedation and Reducing Neurological Dysfunction and Mortality in Septic Patients with Acute Respiratory Failure trial. Crit Care Resusc. 2020 Mar;22(1):63-71. doi: 10.51893/2020.1.oa7. PMID 32102644

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 438 participants signed consent and were enrolled in the clinical trial. 16 participants screen-failed and were ineligible for randomization. 422 participants were randomized and assigned to an arm/treatment group
Groups:
- Dexmedetomidine: Route and Concentration. The study drug will be administered intravenously (IV) by continuous infusion at concentrations of 5 mcg/mL dexmedetomidine. Patients will only receive study drug while in the ICU and on mechanical ventilation, and thus will be monitored with continuous telemetry as per usual ICU practice.
  Dosing Range. Study drug dose will be titrated in a double-blind manner according to clinical effect to achieve a "goal" or "target" Richmond Agitation Sedation Score set by the managing clinical team. For patients in the dexmedetomidine group, dose will range from 0.15-1.5 mcg/kg/hr.
  Dexmedetomidine: For patients in the dexmedetomidine group, dose will range from 0.15-1.5 mcg/kg/hr. For example, a 70 kg patient would receive 10.5 mL of study drug per hour, which would provide 0.75 mcg/kg/hr of dexmedetomidine. This dose range have been selected after literature review and discussions with critical care practitioners, investigational pharmacists, and the MENDS2 study steering committee.
- Propofol: Route and Concentration. The study drug will be administered intravenously (IV) by continuous infusion at concentrations of 10 mg/mL propofol. Patients will only receive study drug while in the ICU and on mechanical ventilation, and thus will be monitored with continuous telemetry as per usual ICU practice.
  Dosing Range. Study drug dose will be titrated in a double-blind manner according to clinical effect to achieve a "goal" or "target" Richmond Agitation Sedation Score set by the managing clinical team. For patients in the propofol group, dose will range from 5-50 mcg/kg/min.
  Propofol: For patients in the propofol group, dose will range from 5-50 mcg/kg/min. For example, a 70 kg patient would receive 10.5 mL of study drug per hour, which would provide 25 mcg/kg/min of propofol. This dose range has been selected after literature review and discussions with critical care practitioners, investigational pharmacists, and the MENDS2 study steering committee.
Period: Overall Study
Arm/Group | Dexmedetomidine | Propofol
Started | 214 (Underwent randomization and received study drug) | 208 (Underwent randomization and received study drug)
Discharged From Hospital and Eligible for Follow-up | 140 | 147
Completed (Alive and completed 6 mos follow-up) | 108 (97% of those eligible (alive and who did not withdraw)) | 101 (91% of those eligible (alive and who did not withdraw))
Not Completed | 106 | 107
Not completed — Death | 89 | 86
Not completed — Withdrawal by Subject | 10 | 8
Not completed — Lost to Follow-up | 3 | 10
Not completed — Did not speak English required for neurospychological testing | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Propofol | Total
Number analyzed (Participants) | 214 | 208 | 422
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [48 to 68] | 60 [50 to 68] | 60 [50 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 88 | 181
  Male | 121 | 120 | 241
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 18 | 30
  Not Hispanic or Latino | 202 | 190 | 392
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 23 | 38
  White | 188 | 177 | 365
  More than one race | 11 | 8 | 19
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 214 | 208 | 422
Informant Questionnaire on Cognitive Decline (IQCODE) Short Form [Median (Inter-Quartile Range); unit: units on a scale] — The Informant Questionnaire on Cognitive Decline (IQCODE) Short Form is a 16 question self-reported measure of cognitive functioning evaluating the degree of decline from baseline. Surrogates in the study must know participant for at least 10 years. Each question includes the prompt, "Compared to 10 years ago how is the patient faring now"? Questions range in score from 1 to 5, with a minimum total survey score of 16 and maximum of 80. An average question score of 3 means the subject is rated as 'no change'. An average score of 4 means 'a bit worse', and an average score of 5 is 'much worse'.
  units on a scale | 3.06 [3 to 3.23] | 3 [3 to 3.25] | 3 [3 to 3.25]
Charlson Comorbities index score [Median (Inter-Quartile Range); unit: units on a scale] — The Charlson Comorbidity Index categorizes comorbidities of participants based on International Classification of Diseases (ICD) diagnosis codes found in administrative data (e.g., hospital records). Each comorbidity category has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use. The sum of all the weights results in a single comorbidity index score for participants ranging from 0 to 37. A score of zero indicates no comorbidities. The higher the score, the more likely the predicted outcome will result in mortality or higher resource use.
  units on a scale | 2 [1 to 4] | 2 [1 to 4] | 2 [1 to 4]
Sequential Organ Failure Assessment (SOFA) score at enrollment [Median (Inter-Quartile Range); unit: units on a scale] — The Sequential Organ Failure Assessment numerically quantifies the number and severity of failed organs. The minimum score is 0, the maximum score is 24, with higher scores indicating higher likelihood of worse outcome
  units on a scale | 10 [8 to 13] | 10 [8 to 12] | 10 [8 to 13]
Infection confirmed by culture [Count of Participants; unit: Participants] | 146 | 132 | 278

OUTCOME MEASURES:

1. Primary Outcome: Delirium/Coma Free Days (DCFDs)
Description: The analysis of DCFDs will be conducted using Intention-to-Treat (ITT) population, defined as all patients who were randomized and received study drug. We chose a 14 day evaluation period for delirium, because it represents the best balance of gaining valuable clinical information, while maximizing resource utilization, given the average study drug infusion to be 7 days and maximum duration to be 14 days. Thus our follow-up period will cover 7 additional days of delirium monitoring after the study drug is stopped in the majority of our patients.
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 214 | 208
days | 8 [1 to 12.8] | 7.5 [1.8 to 11.2]

2. Secondary Outcome: Ventilator-free Days (VFDs)
Description: Ventilator-free days (VFDs), i.e., days alive and free of mechanical ventilation (MV) at 28 days. This endpoint has been used by the National Heart, Lung, and Blood Institute (NHLBI) ARDSNet in numerous critical care trials examining ICU populations.
Time Frame: 28 Days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 214 | 208
days | 20.9 [0 to 26.1] | 19.9 [4.2 to 24.9]

3. Secondary Outcome: Death at 90 Days
Description: That sedation of mechanically ventilated severely septic patients with an alpha2 agonist (dexmedetomidine) rather than a GABAergic agent (propofol) will improve 90-day survival of ICU patients.
Time Frame: 1 through 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 214 | 208
Participants | 81 | 82

4. Secondary Outcome: Cognitive Function Utilizing the Telephone Interview for Cognitive Status Total (TICS-T)
Description: The Telephone Interview for Cognitive Status is a standardized test of cognitive functioning that monitors changes in cognitive functioning over time. The TICS-T consists 11 items including wordlist memory, orientation, attention, repetition, conceptual knowledge and nonverbal praxis. Age-adjusted total scores on the TICS-T range from 0 to 100 with a mean of 50+/-10; lower scores indicate worse cognition, and a score of 35 or less indicates cognitive impairment.
Time Frame: 6 months after randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 214 | 208
score on a scale | 39 [28 to 48] | 38 [30 to 46]

ADVERSE EVENTS:
Time Frame: Up to 30 days since enrollment of discharge whichever came first
Description: Safety endpoints were collected as outcomes, and given the high rates of metabolic and organ dysfunctions, these have been reported separately in the manuscript. Adverse events excluding those and attributable to the study were not found
Arm/Group | Dexmedetomidine | Propofol
All-Cause Mortality (participants affected / at risk) | 89/214 | 86/208
Serious Adverse Events (participants affected / at risk) | 0/214 | 0/208
Other Adverse Events (participants affected / at risk) | 0/214 | 0/208

LIMITATIONS AND CAVEATS:
Sample size readjusted to 420 with approval from NIH and DSMB

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT01739933/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT01739933/SAP_002.pdf